CLINICAL TRIAL: NCT01029951
Title: Neck Pain Comparative Study
Brief Title: Relative Effectiveness and Adverse Effects of Cervical Manipulation, Mobilisation and the Activator Instrument in Patients With Sub-acute Non-specific Neck Pain: a Pragmatic Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglo-European College of Chiropractic (Other)
Collaborators: European Chiropractors Union (Unknown); National Institute for Chiropractic Research (Unknown)
Responsible Party: Hugh Gemmell Principal Lecturer, Anglo-European College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A.06-2
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2006-07

CONDITIONS: Neck Pain
Keywords: Chiropractic; osteopathic physicians; manipulation; neck pain; adverse effects; randomized clinical trial; Subacute non-specific neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: manipulation
Procedure: Mobilisation
Device: Activator instrument

SUMMARY:
The primary purpose of this study was to compare the relative effectiveness of cervical manipulation, mobilisation and the Activator instrument in the treatment of subacute non-specific neck pain. The secondary purpose was to describe any adverse effects of these treatments.

DETAILED DESCRIPTION:
Neck pain is a common disorder. About 70% of adults will experience neck pain during their lifetime. After low back pain, neck pain is the most common reason patients give for seeking chiropractic care, and the second most common reason for the use of spinal manipulation. Usually, the underlying cause of neck pain is non-specific and cannot be related to a particular pathology as a cause of the presenting symptoms. Due to the uncertainty of the results obtained in the limited number of studies of manipulation and mobilisation for neck pain, further studies are needed to compare the different therapies available for neck pain. Participants in the study were treated as they would normally be with the exception of the type of spinal manipulation. There were three groups: a manipulation group, a mobilisation group, and an Activator instrument group.

ELIGIBILITY:
Inclusion Criteria:

* age 18-64 years; a new or recurrent episode of neck pain present for more than 4 weeks, but no longer than 12 weeks;
* neck pain that could extend to the shoulder region or upper extremities, and be accompanied by headache, but neck pain was more painful;
* the patient agreed not to take medication or receive other treatment for neck pain during the course of the study (paracetamol 500 mg 4 times a day was allowed as rescue medication);
* and a baseline pain level of at least 4 on the 11-point numerical rating scale.

Exclusion Criteria:

* Exclusion criteria were treatment with any of the interventions during 6 months prior to recruitment to the study; specific neck pain due to fracture, neoplasm, infection, inflammatory arthropathy, radiculopathy or myelopathy;
* factors contraindicating manipulation, such as blood coagulation disorders, long-term use of corticosteroids, anticoagulant medications, history of neck surgery, stroke or transient ischaemic attacks; plans to relocate;
* inability to read or understand English;
* and third-party liability or workers' compensation claims.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change | end of treatment, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Numerical rating scale for pain | end of treatment, 3 months, 6 months, and 12 months
Bournemouth Questionnaire | end of treatment, 3 months, 6 months, and 12 months
Adverse effects to treatment | end of treatment
SF-36 version 2 | end of treatment, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A Gemmell, DC. EdD, Principal Investigator — Asociación Española contra el Cáncer
Locations (1):
- Anglo-European College of Chiropractic Out Patient Clinic, Bournemouth, Dorset, United Kingdom